CLINICAL TRIAL: NCT03390023
Title: Finding Opportunities for Clinical Care and Trial Participation Among Underrepresented Samples: An Administrative Supplement to the ADORE Trial
Brief Title: Finding Opportunities for Clinical Care and Trial Participation Among Underrepresented Samples
Acronym: ADORE FOCUS
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: STUDY00141699; 3R01HD083292-02S1 (NIH)
Record Dates: First submitted 2017-12-26; First posted 2018-01-04 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Pregnancy Related
Keywords: Prenatal Care; Barriers; Clinical Trials
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hispanic Women: Hispanic women who have been pregnant within the past 5 years.
  Interventions: Behavioral: Focus Group
- Close Family Member: Close family member of participants in Group 1 - Hispanic Women.
  Interventions: Behavioral: Focus Group

INTERVENTIONS:
Behavioral: Focus Group — Groups will last 60 to 90 minutes. Focus groups will be moderated by KUMC Juntos staff who are formally trained to conduct focus groups. General topics to be covered in focus groups include: attitudes, preferences and knowledge about prenatal care, clinical trial participation, and nutritional supplement use. Focus groups will be conducted in Spanish.

SUMMARY:
Focus groups for Hispanic women who are pregnant and their close family members to assess attitudes, barriers and cultural beliefs involved in participation in clinical trials

DETAILED DESCRIPTION:
This is a qualitative study conducted with Hispanic pregnant women and their families. Focus groups for Hispanic pregnant women will run concurrent to groups for their close family member, but in separate rooms. Each focus group session of approximately 8-10 participants is expected to last 60-90 minutes and will be led by an experienced moderator who is fluent in Spanish. All discussions will be audio taped and will be kept confidential. Information learned will be used to refine clinical trial procedures and ensure our model of recruitment and retention in the parent ADORE Trial (NCT02626299) is culturally and linguistically acceptable and feasible.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic women between the ages of 18.0-49.99 yrs old who have been pregnant within the past 5 years OR a close family member
* Speak and understand Spanish

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Focus group participants will be identified both from community health fairs, community events and from local obstetrics and gynecology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Exploratory results from focus groups: access to and attitudes towards prenatal care | 1 year
  Qualitative description of barriers to access in prenatal care
Exploratory results from focus groups: access to and attitudes towards clinical trials | 1 year
  Qualitative description of perceptions and beliefs regarding clinical trial research

CONTACTS AND LOCATIONS:
Overall Officials: Susan Carlson, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- See also: Main Study Clinicaltrials.gov Record: Assessment of DHA On Reducing Early Preterm Birth (ADORE) — https://clinicaltrials.gov/ct2/show/NCT02626299